CLINICAL TRIAL: NCT03660631
Title: Dissemination of the Cardiovascular Risk Service
Acronym: CVRSLive
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korey Kennelty (Other)
Responsible Party: Sponsor-Investigator, Korey Kennelty, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201710812
Record Dates: First submitted 2018-08-20; First posted 2018-09-06 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hypertension; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Patient subjects will participate in their office's randomization group (intervention or control) for the 1st 12 months of their participation. After 12 months, each patient subject in the control group will receive the study intervention for months 13-24. Patient subjects in the intervention will be followed by study pharmacists during months 13-24.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVRS Early Intervention (Experimental): Patients participating in intervention offices will receive the pharmacist-led CVRS intervention for 12 months.
  Interventions: Behavioral: CVRS Intervention
- CVRS Delayed Intervention (Other): Patients participating in control site offices will not have any contact with the CVRS pharmacist for the first 12 months of their participation in the study. They will receive the study intervention during months 13-24.
  Interventions: Behavioral: CVRS Intervention

INTERVENTIONS:
Behavioral: CVRS Intervention — 1. Evaluate gaps in therapy
  2. Contact patients regularly by email, phone and/or text message
  3. Assess and counsel for medication adherence, side effects, life-style behaviors
  4. Develop an action plan and send recommendations to provider

SUMMARY:
The objective of this study is to evaluate the implementation of of a remote, pharmacist-led cardiovascular risk service (CVRS) in 12 large, organizationally and culturally diverse hospitals and health-systems, many with high proportions of minority and underserved patients.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) causes 2,200 deaths in Americans every day with one death every 39 seconds. Yet effective implementation of research-based interventions that reduce CVD-related illness and death remains a substantial challenge. The objective of this study is to test the scalability of a pharmacist-led, remote CVD risk and prevention services model in large, organizationally and culturally diverse hospitals and health-systems, many with high proportions of minority and underserved patients, using a pragmatic cluster-randomized design. This service is called the Cardiovascular Risk Service (CVRS). There are limited data on the barriers and facilitators of implementation to enhance the CVRS in these types of diverse, complex health-systems. Therefore, scaling up our effective, innovative team-based intervention will require an assessment of barriers and facilitators to CVRS adoption, implementation, and maintenance. Our central hypothesis is that barriers and facilitators to CVRS implementation will vary across diverse primary care offices. We will use mixed methods including interviews, observations, and an innovative physician-pharmacist collaboration survey we developed to predict implementation of pharmacy-based services. The rationale for this proposed study is that overcoming barriers to implementation of a novel strategy to improve secondary prevention of CVD will lead to innovative strategies for broader adoption by health systems throughout the US.

ELIGIBILITY:
Inclusion Criteria:

* Patient Subjects:

  * English or Spanish speaking
  * Seen in the clinic at least once in the previous 12 months
  * Currently has one of the following diseases:

    1. Diabetes with HA1c 9.0% or greater and/or
    2. Hypertension (uncomplicated) with systolic blood pressure 150 mm Hg or greater

Exclusion Criteria:

* Inability to give consent
* Nursing home residence
* No telephone

  * Additional patient subject exclusions:
* Cancer with a life expectancy less than 24 months
* Pregnancy
* Diagnosis of dementia
* Plans to terminate care from the clinic within 24 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Factors influencing intervention implementation fidelity | 12 months following the start of the intervention at each site
  Themes will be identified through interviews with key individuals involved in implementation of study intervention. Data from interviews will be analyzed using ATLAS ti to determine frequency and density of themes identified in interviews.
Effect of physician/pharmacist collaboration on implementation fidelity | 12 months following the start of the intervention at each site
  Development of implementation fidelity measures and adherence to fidelity measures

SECONDARY OUTCOMES:
Adherence to guidelines for primary and secondary prevention of cardiovascular disease | 12 months after the start of the intervention for each subject
  The percent of select Guideline Advantage criteria met by subjects in the Early Intervention arm versus the Delayed Intervention arm
Reach and adoption of intervention | 12 months following the start of the intervention at each site
  Proportion of patients and providers participating who were approached
Development of payment contracts | 36 months following the start of recruitment
  Create a template for payment contracts between clinical sites and the CVRS
Development of payment contracts | 36 months following the start of recruitment
  The number of clinical sites that successfully negotiate payment contracts with the CVRS

CONTACTS AND LOCATIONS:
Overall Officials: Korey Kennelty, PharmD, Principal Investigator — University of Iowa
Locations (14):
- United States (14):
  - Idaho State University, Pocatello, Idaho
  - University of Illinois at Chicago: Mile Square Health Center, Chicago, Illinois
  - Carle Foundation Hospital, Mahomet, Illinois
  - Carle Foundation Hospital, Rantoul, Illinois
  - Genesis Family Medical Center, Davenport, Iowa
  - University of Iowa, Iowa City, Iowa
  - UIHC River Crossing, Riverside, Iowa
  - Siouxland Family Medicine Center, Sioux City, Iowa
  - Northeast Iowa Family Practice Center, Waterloo, Iowa
  - Henry Ford Health System: Harbortown, Detroit, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Texas Tech University Health Science Center, Amarillo, Texas
  - Community Health Center of Snohomish County, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
1. Provide de-identified SAS datasets in transport format with the protocol, data dictionaries user manual . A data sharing agreement will be required.
  2. Share data with all participating sites and place study links and information on PBRN website136
  3. Present results to other PBRNs through AHRQ meetings.
  4. Post the development and results on the .213 PRagmatic-Explanatory Continuum Indicator Summary
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months following the start of the study intervention.

REFERENCES:
- [Derived] Kennelty KA, Engblom NJ, Carter BL, Hollingworth L, Levy BT, Finkelstein RJ, Parker CP, Xu Y, Jackson KL, Dawson JD, Dorsey KK. Dissemination of a telehealth cardiovascular risk service: The CVRS live protocol. Contemp Clin Trials. 2021 Mar;102:106282. doi: 10.1016/j.cct.2021.106282. Epub 2021 Jan 12. PMID 33444781